CLINICAL TRIAL: NCT06314568
Title: Radiochemotherapy Treatment Followed by Interventional Radiotherapy in Patients Affected by Vagina Carcinoma Multi-centric Prospective Observational Study Trimodal Definitive Invasive Vaginal Carcinoma Treatment
Brief Title: Radiochemotherapy and Interventional Radiotherapy in Vaginal Cancer
Acronym: TRIDENT
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6350
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Vaginal Cancer
MeSH Terms: conditions — Vaginal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with vaginal cancer: Patients affected by vaginal cancer
  Interventions: Radiation: Radiochemotherapy plus interventional radiotherapy

INTERVENTIONS:
Radiation: Radiochemotherapy plus interventional radiotherapy — All patients with vaginal cancer will undergo radiochemotherapy (45 Gy on pelvis and tumor in association with cisplatinum) plus interventional radiotherapy (28 Gy on residual disease) with exclusive intent

SUMMARY:
Prospective observational multicenter study, aimed at evaluating the effectiveness on local control and cancer-specific survival of radiochemotherapy followed by interventional radiotherapy in patients affected by vaginal cancer

DETAILED DESCRIPTION:
Prospective observational multicenter study, aimed at evaluating the effectiveness on local control and cancer-specific survival of radiochemotherapy (45Gy on pelvis and tumor plus chemotherapy with cisplatinum) followed by interventional radiotherapy (28Gy on residual tumor) in patients affected by vaginal cancer

ELIGIBILITY:
Inclusion Criteria:

* Age more than18 years old
* Performance status 0,1
* Hystological diagnosis of squamous vaginal cancer
* HPV, p16, p53 status
* Stage I, II, III and IV (AJCC 2018th version)
* Stadiation with magnetic resonance and positron emission tomography
* Informed consensus

Exclusion Criteria:

* Age inferior 18 years old
* Performance status more than 2
* Previous cancer in the last ten years
* Previous radiation treatment in the region of interest
* Presence of pathologies that contraindicate radiotherapy treatment (genetic syndromes of hyper-radiosensitivity, ulcerative colitis, diverticulitis in the acute phase, severe diverticulosis, chronic pelvic inflammation)
* Presence of internal pathologies that contraindicate chemotherapy or radio-chemotherapy treatment (severe liver disease, heart disease, renal failure, etc.)
* Presence of distant metastases in sites other than the pelvic lymph nodes
* Any significant medical condition that in the opinion of the investigator may interfere with the patient's optimal participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with vaginal cancer that after first consultation will undergo to radiochemotherapy and interventional radiotherapy
Sampling Method: Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Local Control | 6 months
  Local control, the Cox regression model and multivariable logistic analysis will be used to analyze the role of clinical-pathological parameters as prognostic and predictive factors of pathological response to treatment

SECONDARY OUTCOMES:
Cancer specific overall survival | 6 months
  The Cox regression model and multivariable logistic analysis will be used to analyze the role of clinical-pathological parameters as prognostic and predictive factors of pathological response to treatment
Toxicities | 6 months
  The safety and tolerability profile of the treatment will be defined by the frequency and severity of adverse reactions as well as their possible correlation with the treatment received.
Overall survivall | 6 months
  The Cox regression model and multivariable logistic analysis will be used to analyze the role of clinical-pathological parameters as prognostic and predictive factors of pathological response to treatment
Disease free survivall | 6 months
  The Cox regression model and multivariable logistic analysis will be used to analyze the role of clinical-pathological parameters as prognostic and predictive factors of pathological response to treatment
Metastasis free survival | 6 months
  The Cox regression model and multivariable logistic analysis will be used to analyze the role of clinical-pathological parameters as prognostic and predictive factors of pathological response to treatment
Changes in quality of life over time | 6 months
  Anova for repeated measures or the corresponding non-parametric Friedman test will be used to identify changes in quality of life over time.

CONTACTS AND LOCATIONS:
Overall Officials: VALENTINA LANCELLOTTA, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy